CLINICAL TRIAL: NCT01279746
Title: The Diagnosis of Occult Deep Vein Thrombosis of the Lower Extremities in Patients Presenting With Hypoxia
Status: Completed | Type: Observational
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Sponsor
Other Study IDs: 0003-10-EMC
Record Dates: First submitted 2010-11-23; First posted 2011-01-19 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: Hypoxia
Keywords: DVT Ultrasound compression Hypoxia Pulmonary Emboli; Occult DVT in hypoxic patients
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ultrasond compression of deep veins
  Interventions: Device: Ultrasound compression of femoral and popliteal veins

INTERVENTIONS:
Device: Ultrasound compression of femoral and popliteal veins — Bedside ultrasound compression of femoral and popliteal veins.

SUMMARY:
The purpose of this study is to prove that bedside Ultrasound Compression is a useful screening tool for the diagnosis of occult deep vein thrombosis in patients presenting to the emergency room with hypoxia.

DETAILED DESCRIPTION:
It is known that 30% of deep vein thrombosis of the extremities is belived to be the precedend of pulmonary emboli; an often fatal disease. It is known that DVT (deep vein thrombosis is often occult.

It is also known that pulmonary embolism is often difficult to diagnose and is often missed especialy in patients with chronic illnesses such as COPD and CHF.

Venous compression ultrsound is an exam that can be preformed bedside. It is preformed by placing a vascular ultrasound transducer on the femoral vein and popliteal and checking its compressibility. If DVT is present in the femoral or popliteal veins the veins will be noncompressible. It has been shown that US compression for DVT can be preformed by physicians in the ER with accuracy and speed.

Presently US compression is not a tool used for detection of occult DVT in the ER. I wish to explore the usefullness of compression US of the lower extremities as a screening tool for DVT In the hypoxic patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting to the Emergency room
* 18 years or older, saturation 94% and under on room air.

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with saturation under 94% room air
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-04; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - HaEmek Medical Center, Afula, Israel
  - HaEmek Medical Center, Afula